CLINICAL TRIAL: NCT03621202
Title: A Clinical Study to Evaluate the Safety and Accuracy of the Saranas Early Bird Bleed Monitoring System for the Detection of Endovascular Procedure Related Bleeding Events
Brief Title: Safety and Accuracy of the Saranas EBBMS for the Detection of Endovascular Procedure Related Bleeding Events
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saranas, Inc. (Industry)
Collaborators: Proxima CRO (Industry); Medical Metrics Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PVP004
Record Dates: First submitted 2018-07-30; First posted 2018-08-08 (Actual); Results first posted 2020-12-28 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Endovascular Procedures
Keywords: large bore; femoral access; internal bleeding; retroperitoneal hematoma; bleeding complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Saranas Early Bird Bleed Monitoring System (EBBMS) (Experimental)
  Interventions: Device: Saranas Early Bird Bleed Monitoring System (EBBMS)

INTERVENTIONS:
Device: Saranas Early Bird Bleed Monitoring System (EBBMS) — Participants will undergo their planned endovascular procedure with monitoring for internal bleeding using the Saranas EBBMS.

SUMMARY:
To evaluate the safety and accuracy of the Saranas EBBMS for the detection of access site related internal bleeding events during large-bore endovascular procedures.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Willing and capable to sign an Informed Consent form
* Planned endovascular procedure such as trans-femoral transcatheter aortic valve replacement (TAVR), balloon aortic valvuloplasty, percutaneous coronary intervention, complex or high-risk percutaneous coronary intervention requiring hemodynamic support device (Impella 2.5, Impella CP, and ECMO), endovascular aortic repair (EVAR), any other endovascular procedures requiring arterial or venous access or surgical insertion of hemodynamic support

Exclusion Criteria:

* Subject is participating, or planning to participate in a clinical trial or study of an investigational product that may influence the data collected for this investigation
* Inability to access artery or vein for the endovascular procedure
* Current active bleeding
* Pre-procedural conditions precluding the realization of a post-procedural CT scan
* Pregnancy
* Mental disability or any other lack of fitness, in the Investigator's opinion, to preclude subject's participation in or ability to complete the study as planned

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Genereux, M.D., Principal Investigator — Gagnon Cardiovascular Institute, Morristown Medical Center
Locations (5):
- United States (5):
  - North Florida Regional Medical Center, Gainesville, Florida
  - Morristown Medical Center, Morristown, New Jersey
  - Columbia University Medical Center, New York, New York
  - Houston Methodist Hospital, Houston, Texas
  - Texas Heart Institute, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nguyen CT, Lee E, Luo H, Siegel RJ. Echocardiographic guidance for diagnostic and therapeutic percutaneous procedures. Cardiovasc Diagn Ther. 2011 Dec;1(1):11-36. doi: 10.3978/j.issn.2223-3652.2011.09.02. PMID 24282682
- [Background] Roger VL, Go AS, Lloyd-Jones DM, Adams RJ, Berry JD, Brown TM, Carnethon MR, Dai S, de Simone G, Ford ES, Fox CS, Fullerton HJ, Gillespie C, Greenlund KJ, Hailpern SM, Heit JA, Ho PM, Howard VJ, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Makuc DM, Marcus GM, Marelli A, Matchar DB, McDermott MM, Meigs JB, Moy CS, Mozaffarian D, Mussolino ME, Nichol G, Paynter NP, Rosamond WD, Sorlie PD, Stafford RS, Turan TN, Turner MB, Wong ND, Wylie-Rosett J; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2011 update: a report from the American Heart Association. Circulation. 2011 Feb 1;123(4):e18-e209. doi: 10.1161/CIR.0b013e3182009701. Epub 2010 Dec 15. PMID 21160056
- [Background] SELDINGER SI. Catheter replacement of the needle in percutaneous arteriography; a new technique. Acta Radiol (Stockh). 1953 May;39(5):368-76. doi: 10.3109/00016925309136722. No abstract available. PMID 13057644
- [Background] Babu SC, Piccorelli GO, Shah PM, Stein JH, Clauss RH. Incidence and results of arterial complications among 16,350 patients undergoing cardiac catheterization. J Vasc Surg. 1989 Aug;10(2):113-6. doi: 10.1067/mva.1989.0100113. PMID 2788227
- [Background] Chandrasekar B, Doucet S, Bilodeau L, Crepeau J, deGuise P, Gregoire J, Gallo R, Cote G, Bonan R, Joyal M, Gosselin G, Tanguay JF, Dyrda I, Bois M, Pasternac A. Complications of cardiac catheterization in the current era: a single-center experience. Catheter Cardiovasc Interv. 2001 Mar;52(3):289-95. doi: 10.1002/ccd.1067. PMID 11246238
- [Background] Kinnaird TD, Stabile E, Mintz GS, Lee CW, Canos DA, Gevorkian N, Pinnow EE, Kent KM, Pichard AD, Satler LF, Weissman NJ, Lindsay J, Fuchs S. Incidence, predictors, and prognostic implications of bleeding and blood transfusion following percutaneous coronary interventions. Am J Cardiol. 2003 Oct 15;92(8):930-5. doi: 10.1016/s0002-9149(03)00972-x. PMID 14556868
- [Background] Yatskar L, Selzer F, Feit F, Cohen HA, Jacobs AK, Williams DO, Slater J. Access site hematoma requiring blood transfusion predicts mortality in patients undergoing percutaneous coronary intervention: data from the National Heart, Lung, and Blood Institute Dynamic Registry. Catheter Cardiovasc Interv. 2007 Jun 1;69(7):961-6. doi: 10.1002/ccd.21087. PMID 17421023
- [Background] Moscucci M, Fox KA, Cannon CP, Klein W, Lopez-Sendon J, Montalescot G, White K, Goldberg RJ. Predictors of major bleeding in acute coronary syndromes: the Global Registry of Acute Coronary Events (GRACE). Eur Heart J. 2003 Oct;24(20):1815-23. doi: 10.1016/s0195-668x(03)00485-8. PMID 14563340
- [Background] Crudu V, Blankenship J, Berger P, Scott T, Skelding K. Complications related to access site after percutaneous coronary interventions: are the adverse events underreported? Catheter Cardiovasc Interv. 2011 Apr 1;77(5):643-7. doi: 10.1002/ccd.22759. Epub 2011 Mar 8. PMID 20824761
- [Background] Sherev DA, Shaw RE, Brent BN. Angiographic predictors of femoral access site complications: implication for planned percutaneous coronary intervention. Catheter Cardiovasc Interv. 2005 Jun;65(2):196-202. doi: 10.1002/ccd.20354. PMID 15895402
- [Background] Kent KC, Moscucci M, Mansour KA, DiMattia S, Gallagher S, Kuntz R, Skillman JJ. Retroperitoneal hematoma after cardiac catheterization: prevalence, risk factors, and optimal management. J Vasc Surg. 1994 Dec;20(6):905-10; discussion 910-3. doi: 10.1016/0741-5214(94)90227-5. PMID 7990185
- [Background] Fruhwirth J, Pascher O, Hauser H, Amann W. [Local vascular complications after iatrogenic femoral artery puncture]. Wien Klin Wochenschr. 1996;108(7):196-200. German. PMID 8677663
- [Background] Berry C, Kelly J, Cobbe SM, Eteiba H. Comparison of femoral bleeding complications after coronary angiography versus percutaneous coronary intervention. Am J Cardiol. 2004 Aug 1;94(3):361-3. doi: 10.1016/j.amjcard.2004.04.036. PMID 15276106
- [Background] Khoury M, Batra S, Berg R, Rama K, Kozul V. Influence of arterial access sites and interventional procedures on vascular complications after cardiac catheterizations. Am J Surg. 1992 Sep;164(3):205-9. doi: 10.1016/s0002-9610(05)81071-2. PMID 1415915

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Saranas Early Bird Bleed Monitoring System (EBBMS)
Started | 66
Completed | 60
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Saranas Early Bird Bleed Monitoring System (EBBMS)
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 76 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 57
  More than one race | 0
  Unknown or Not Reported | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28 (6)
Hypertension [Count of Participants; unit: Participants] | 37
Diabetes [Count of Participants; unit: Participants] | 25
Atrial Fibrillation [Count of Participants; unit: Participants] | 17
Renal Insufficiency [Count of Participants; unit: Participants] | 7

OUTCOME MEASURES:

1. Primary Outcome: Cohen's Kappa Coefficient (κ)
Description: Statistic measures concordance in detecting bleeds between the Saranas EBBMS and post-procedural CT. Cohen suggested the Kappa result be interpreted as follows: values ≤ 0 as indicating no agreement and 0.01-0.20 as none to slight, 0.21-0.40 as fair, 0.41- 0.60 as moderate, 0.61-0.80 as substantial, and 0.81-1.00 as almost perfect agreement.
Time Frame: Up to 8 hours post procedure
Measure: Number; unit: proportion of agreement
Arm/Group | Saranas Early Bird Bleed Monitoring System (EBBMS)
Number analyzed (Participants) | 60
proportion of agreement | 0.84

2. Secondary Outcome: Device Sensitivity in Bleeding Detection of the Saranas EBBMS as Compared to Post-procedural Computerized Tomography
Description: Sensitivity measures the proportion of positives bleed detection events that are correctly identified by the EBBMS as compared to post-procedural computerized tomography.
Time Frame: Up to 8 hours post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Saranas Early Bird Bleed Monitoring System (EBBMS)
Number analyzed (Participants) | 60
Participants | 60
Statistical Analysis 1: Comparison: Saranas Early Bird Bleed Monitoring System (EBBMS); Test type: Other; The EBBMS sensitivity was 100%

3. Secondary Outcome: Device Specificity in Bleeding Detection of the Saranas EBBMS as Compared to Post-procedural Computerized Tomography
Description: Specificity relates to the EBBMS' ability to correctly reject non-bleeding events as compared to post-procedural computerized tomography.
Time Frame: Up to 8 hours post procedure
Measure: Number; unit: Percentage
Arm/Group | Saranas Early Bird Bleed Monitoring System (EBBMS)
Number analyzed (Participants) | 60
Percentage | 75
Statistical Analysis 1: Comparison: Saranas Early Bird Bleed Monitoring System (EBBMS); Test type: Other; The EBBMS specificity was 75%

ADVERSE EVENTS:
Time Frame: 5 months
Arm/Group | Saranas Early Bird Bleed Monitoring System (EBBMS)
All-Cause Mortality (participants affected / at risk) | 2/60
Serious Adverse Events (participants affected / at risk) | 9/60
Other Adverse Events (participants affected / at risk) | 28/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Saranas Early Bird Bleed Monitoring System (EBBMS) (N=60)
Clot on right atrium of tricuspid valve (Cardiac disorders) | 1 (1)
CAD with acute ischemia (Cardiac disorders) | 1 (1)
Symptomatic anemia (General disorders) | 1 (1)
Hypertension/SOB/Fluid overload (General disorders) | 1 (1)
Coronary or RV perforation w cardiac tamponade (Cardiac disorders) | 1 (1)
Prolonged bleeding from left groin (Vascular disorders) | 1 (1)
Pseudoaneurysm (Vascular disorders) | 1 (1)
2:1 High Grade AV Block (Cardiac disorders) | 1 (1)
CVA / Bleed (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Saranas Early Bird Bleed Monitoring System (EBBMS) (N=60)
2:1 High Grade AV Block (Cardiac disorders) | 1 (1)
A-V Fistula (Vascular disorders) | 1 (1)
Blood Loss Anemia (Blood and lymphatic system disorders) | 2 (2)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrial Fib & RVR (Cardiac disorders) | 1 (1)
Back Pain (General disorders) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
CVA (General disorders) | 2 (2)
Delirium (Psychiatric disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
EKG Changes (Cardiac disorders) | 1 (1)
Elevated Creatinine (Renal and urinary disorders) | 1 (1)
Fever 100.8 Unknown Source (General disorders) | 1 (1)
Generalized Pain (General disorders) | 1 (1)
Gron Pain (General disorders) | 3 (3)
Headache (General disorders) | 1 (1)
Hematemesis (Gastrointestinal disorders) | 1 (1)
Hyperkalemia (Renal and urinary disorders) | 1 (1)
Hypertension (General disorders) | 1 (1)
Hypotension (General disorders) | 1 (1)
New LBBB (Cardiac disorders) | 5 (5)
Leg Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Leukocystosis (General disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
New Prolonged P-R Interval (Cardiac disorders) | 1 (1)
Polyarthralgias (Musculoskeletal and connective tissue disorders) | 1 (1)
Pseudoaneurysm (Vascular disorders) | 1 (1)
R Temporal Artery Bleed (Vascular disorders) | 1 (1)
Right Arm Pain - Generalized (General disorders) | 1 (1)
Right Upper Extremity Swelling (General disorders) | 1 (1)
SOB & Fluid Retention (General disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 1 (1)
Worsening Heart Failure (Cardiac disorders) | 2 (2)
Worsening Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-04): https://cdn.clinicaltrials.gov/large-docs/02/NCT03621202/Prot_SAP_000.pdf
  • Informed Consent Form (2018-05-04): https://cdn.clinicaltrials.gov/large-docs/02/NCT03621202/ICF_002.pdf